CLINICAL TRIAL: NCT01355341
Title: A Phase II, 28 Week, Randomized, Double- Blind, Placebo- Controlled, Parallel Group Study to Evaluate the Safety and Efficacy of 'Herbmed Plus' an Ayurvedic Formulation in Patients With Renal Calculi
Brief Title: Safety and Efficacy of Herbmed Plus in Patients withRenal Calculi
Acronym: HerbmedPlus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amai Charitable Trust (Other)
Responsible Party: AMAI CHARITABLE TRUST'S ACE HOSPITAL PUNE, AMAI CHARITABLE TRUST
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACE/HMP-01
Record Dates: First submitted 2011-05-16; First posted 2011-05-18 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2011-05

CONDITIONS: RENAL CALCULI
Keywords: RENAL CALCULI HERBMED PLUS
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- HERBMED PLUS (Experimental): Herbal formulation of four constituents i.e.Varuna,Yav,Aghada,Kadali as per ayurvedic literature.
  Interventions: Drug: HERBMED PLUS

INTERVENTIONS:
Drug: HERBMED PLUS — 500 mg Twice day for 6 month with lunch and dinner.
  Other Names: Herbmed plus is ayurvedic formulation

SUMMARY:
More specifically, the present invention relates to a 'Herbal Preparation' that is useful for

* Treatment of Renal calculi
* Reduction in the stone size & surface area
* The expulsion of stone
* Decreased need of Analgesic(Antiinflammatory Effect)
* Stops the recurrence and reformation of renal

DETAILED DESCRIPTION:
1. Study duration 28 weeks
2. No. of Scheduled visits 8 visits
3. Study product Dose, Group one-:1capsule (of 500 mg) orally twice a day with meals for 24 weeks. Group two-:placebo1capsule (of 500 mg) orally twice a day with meals for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 10-75 years (Both inclusive)
* Patients with Renal calculi, diagnosis confirmed by plain X-ray KUB &/or ultrasound KUB/CT scan Abdomen
* Size of the calculi ranging from 04 mm -09 mm
* Able and willing to give written informed consent and comply with the requirements of the study protocol
* Patients of reproductive potential (males and females) and willing to use a reliable means of contraception (e.g hormonal contraceptive patch, intrauterine device and physical barrier) throughout study participation
* Patients will to cooperate & give consent for the trial& comes for regular follow up.

Exclusion Criteria:

* Patients having acute condition of renal calculi.
* Any systemic disease requiring other medications of surgery for calculus condition.
* Complicated cases of Renal Calculi requiring surgical condition.
* Chronic or current infectious disease such as but not limited to chronic renal infection including active urinary tract infection.Uncontrolled diabetes, hypertension, symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction
* Any other urogenital disorders.
* Liver dysfunction, defined as total bilirubin more then 1.5 the upper limit of Normal, aspartate aminotransferase more then 2.5 upper limit of Normal, or alanine aminotransferase more then 2.5 upper limit of Normal,
* Kidney disease, including serum creatinine level more then 1.5 upper limit of Normal,
* Subjects on herbal supplements for stone disease (plant extracts preparations or herbal medicines etc.) within previous 3 months.
* Participated in another clinical drug trial within 3 months before recruitment.
* Pregnancy or breast feeding
* Evidence of significant uncontrolled concomitant disease which in the Investigator's opinion would preclude patient participation
* Currently active alcohol or drug abuse or history of alcohol or drug abuse within 24 weeks prior to baseline
* Patients with psychiatric illness or other condition that would limit compliance with study requirements
* Patients receiving or has received any investigational drug within 30 days before receiving the first dose of study medication
* Subjects who refuse to sign the informed consent document .

Ages: 10 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of "Herbmed plus"in patients with urinary calculi by assessing the reduction in the stone size & surface area/ or the expulsion of stone | In 210 days

SECONDARY OUTCOMES:
Reduction in the size of stone Reduction in the density of the stone Painless expulsion of the stone/fragments Reduction in pain Consumption of Analgesics | In 210 days

CONTACTS AND LOCATIONS:
Overall Officials: SURESH B PATANKAR, MS.Mch., Principal Investigator — AMAI CHRITABLE TRUST'S ACE HOSPITAL
Locations (1):
- AMAI Charitable Trust's ACE Hospital Pune, Pune, Maharashatra, India